CLINICAL TRIAL: NCT01089049
Title: A Clinical Trial to Assess the Efficacy of a Supplemental Formula Targeting Breast Health in Beneficially Altering Urinary Estrogen Metabolites Levels in Both Pre- and Post-menopausal Women
Brief Title: Effect of a Natural Health Product on Urinary Estrogen Metabolites
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NDI: 136987; NHPD136987 (Other: Natural Health Products Directorate, Health Canada)
Record Dates: First submitted 2010-03-12; First posted 2010-03-18 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Breast Cancer
Keywords: Urinary Estrogen Metabolites; 2-OH Estrone; 16-alpha-OH Estrone; Urinary 2/16a Estrogen Metabolite Ratio
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre-Menopausal (Experimental)
  Interventions: Dietary Supplement: FemMED Breast Health Formula
- Post-Menopausal (Experimental)
  Interventions: Dietary Supplement: FemMED Breast Health Formula

INTERVENTIONS:
Dietary Supplement: FemMED Breast Health Formula — Two capsules daily, with meals. FemMED Breast Health Formula containing lignans.

SUMMARY:
The purpose of this study is to determine if a supplemental formula can beneficially alter the ratio of urinary estrogen metabolites.

DETAILED DESCRIPTION:
The active botanical constituents in femMED Breast Health Formula contain lignans, compounds with anti-estrogenic activity, that have been shown to exert an estrogenic effect during the follicular phase [i.e. when estrogen is low] and an antiestrogenic effect in the luteal phase of a female menstrual cycle. These are plant-derived chemicals that can act as weak mimics of estrogen in the body. Overall these compounds have been found to be helpful in stabilizing the natural cyclical fluctuation of estrogen levels.

The trial will be a double-blind, placebo-controlled parallel study in which 100 subjects will be recruited to one of two arms of the study: one arm will consist of pre-menopausal women; another will consist of post-menopausal women. Each arm of the study will be carried out concurrently and in one phase, with no washout period. The placebo assignment will be randomized within each arm of the study.

Subjects in each arm of the study will follow the same protocol. Urine and blood samples will be collected from each group at both the first and last visit, and subjects will receive a month's supply of treatment or placebo at the first visit, which they will consume on a daily basis until their second lab visit 28 days later. Urine samples will be analyzed for the following estrogen metabolites: 2-OH-estrone and 16-α OH-estrone. Blood samples would be collected and assessed for levels of enterolactone. Pre and post-supplementation results will be assesses for any differences by statistical comparison.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Healthy
* Willing to collect urine samples and to have blood drawn
* Post-menopausal and have not taken hormone replacement therapy (HRT) in the past year (48 subjects)
* Pre-menopausal (48 subjects)

Exclusion Criteria:

* Diagnosed with any major illness(e.g. cancer)
* Diabetes, thyroid disease, atypical hyperplasia, fibrocystic breast disease, family history of ovarian cancer, a history of "migraines with aura"
* Women taking blood thinner or thyroid medication (including warfarin)
* Known allergy to any of the any of the study ingredients
* Pregnancy or lactation
* Regular consumption in the previous 3 months of any other natural health products (NHPs) or pharmaceutical containing ingredients with a similar effect on estrogen metabolism as those included in the femMED Breast Health treatment
* Family history of breast cancer risk
* Post-menopausal women on HRT
* Pre-menopausal women taking hormonal contraceptives (oral contraceptives, the patch etc.)
* All other forms of estrogen, progesterone and/or androgens (i.e. testosterone therapy)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2009-08; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
2-OH Hydroxy Estrone: 16-alpha-OH Estrone | Day 0, Day 28
  2-OHE:16α-OHE1 (2:16 ratio) - 2:16 ratios less than 2.0 indicate increasing long-term risk for breast, cervical, and other estrogen sensitive cancers.
  Urine samples will be analyzed for the following estrogen metabolites: 2-OH-estrone and 16-α OH-estrone.

SECONDARY OUTCOMES:
Enterolactone | Day 0, Day 28
  Enterolactone is a lignan formed by the action of intestinal bacteria on lignan precursors found in plants. For the purpose of this study, enterolactone will serve as an indicator of compliance/dietary intake of lignans.
  Blood samples would be collected and assessed for levels of enterolactone.

CONTACTS AND LOCATIONS:
Overall Officials: Maggie Laidlaw, P.hD, Principal Investigator — Nutrasource Pharmaceutical and Nutraceutical Services, Inc.
Locations (1):
- Nutrasource Diagnostics Inc, Guelph, Ontario, Canada

REFERENCES:
- [Derived] Laidlaw M, Cockerline CA, Sepkovic DW. Effects of a breast-health herbal formula supplement on estrogen metabolism in pre- and post-menopausal women not taking hormonal contraceptives or supplements: a randomized controlled trial. Breast Cancer (Auckl). 2010 Dec 16;4:85-95. doi: 10.4137/BCBCR.S6505. PMID 21234288